CLINICAL TRIAL: NCT07149129
Title: Use of Electromyographic Biofeedback in Upper Limb Rehabilitation After Stroke
Brief Title: Biofeedback After Stroke
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Paraná (Other)
Collaborators: UTFPR (Unknown)
Responsible Party: Principal Investigator, Henrique Cunha Carvalho, PhD., Universidade Federal do Paraná
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 84156424.6.0000.5547; 84156424.6.0000.5547 (Registry Identifier: APPROVAL BY THE ETHICS COMMITTEE - CEP UTFPR)
Record Dates: First submitted 2025-08-14; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: muscle spasticity; stroke; biofeedback; electromyography
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: Sham group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMG Biofeedback - Intervention (Placebo Comparator): This intervention phase will last 30 minutes of training, during which the participant will be encouraged to actively and voluntarily relax their spastic muscles and will receive visual feedback through the software when this occurs. Two modes will be used in the software: the first, called "Recovery", which consists of a game in which the participant is encouraged to contract and relax their muscles in order to guide a rocket in a specific direction to earn points. The second, called "Maestro", in which the participant's objective is to keep the rocket below the specified line while maintaining their muscles relaxed. The participant will perform each mode for 15 minutes, totaling the proposed 30 minutes. There may be a break between each mode if the participant experiences fatigue. Afterward, they will receive standard occupational therapy.
  Interventions: Device: Electromyographic Biofeedback
- EMG Biofeedback - Sham (Sham Comparator): The intervention with the placebo (sham) group will have an identical structure to that of the intervention group, but during the biofeedback phase, the software screen will be a simulation, not corresponding to the patient's muscle activity. The patient will receive occupational therapy as usual, in a manner identical to that of the intervention group after the placebo biofeedback therapy.
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: Electromyographic Biofeedback — This intervention phase will last 30 minutes of training, during which the participant will be encouraged to actively and voluntarily relax their spastic muscles and will receive visual feedback through the software when this occurs. Two modes will be used in the software: the first, called "Recovery", which consists of a game in which the participant is encouraged to contract and relax their muscles in order to guide a rocket in a specific direction to earn points. The second, called "Maestro", in which the participant's objective is to keep the rocket below the specified line while maintaining their muscles relaxed. The participant will perform each mode for 15 minutes, totaling the proposed 30 minutes. There may be a break between each mode if the participant experiences fatigue. Afterward, they will receive standard occupational therapy.
  Arms: EMG Biofeedback - Intervention
Device: Sham (No Treatment) — The intervention with the placebo group will have an identical structure to that of the intervention group, but during the biofeedback phase, the software screen will be a simulation, not corresponding to the patient's muscle activity. The patient will receive occupational therapy as usual, in a manner identical to that of the intervention group after the placebo biofeedback therapy.
  Arms: EMG Biofeedback - Sham

SUMMARY:
Studies show that the use of electromyographic biofeedback combined with other therapies contributes to the reduction of upper limb spasticity after stroke. However, there is a lack of literature regarding the best protocols to use in clinical practice, as well as functional outcomes after this therapy. The objective of this research project will be to investigate the effect of electromyographic biofeedback on spasticity in individuals post-stroke in the sub-acute phase, and its outcomes regarding upper limb function and participation in activities of daily living. The study will be a randomized, triple-blind clinical trial in which the 45 participants will be divided into two groups: the experimental group will receive electromyographic biofeedback combined with functional training, and the control group will receive functional training with placebo biofeedback alone. The study hypothesis is that the use of electromyographic biofeedback contributes to improved functional outcomes and participation in activities of daily living in patients with upper limb spasticity resulting from stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of stroke (imaging tests and a medical report)
* Spasticity with an Ashworth score equal to or less than 3 in the upper limb
* 20-60 years old

Exclusion Criteria:

* Other neurological impairments or trauma-orthopedic deformities in the upper limbs
* botulinum toxin/phenol injections within the previous 5 months
* medications that reduce muscle tone
* aphasia that prevents basic communication
* low vision or low visual acuity that prevents them from viewing the screen.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Ashworth | Ashworth will be applied at pre (baseline), through study completion, an average of 1 month.
  The Ashworth scale will be used to measure the degree of spasticity of the upper limb muscles. The test will be performed manually and the score ranges from zero to four points. The higher the score, the greater the spasticity of the muscle tested.

SECONDARY OUTCOMES:
Upper limb function and participation - The Functional Independence Measure (FIM) | The tests will be applied at pre (baseline), through study completion, an average of 1 month.
  The Functional Independence Measure (FIM) will be used to potentially classify the level of dependence of the subject as: complete (18 to 45 points), moderate independence (46 to 99), and full independence (100 to 126). The lower the subject's score, the more dependent they are. The minimally clinically important difference for this evaluation is 22 points.
Upper limb function and participation - Modified Ashworth scale | The tests will be applied at pre (baseline), through study completion, an average of 1 month.
  The Modified Ashworth scale will be used to measure the degree of spasticity in the upper limb musculature. The score ranges from zero to four points. The higher the score, the greater the spasticity of the tested muscle.
Upper limb function and participation - Motor Activity Log (MAL) | The tests will be applied at pre (baseline), through study completion, an average of 1 month.
  The Motor Activity Log (MAL) measures how much the upper limb is used in daily activities. The average is directly proportional to the quantity and quality of upper limb use. In both scales, the minimally clinically relevant difference is 1.0 points if the paretic limb is not dominant or 1.1 points if the paretic limb is dominant.
Upper limb function and participation - Box and Block Test (BBT) | The tests will be applied at pre (baseline), through study completion, an average of 1 month.
  In the Box and Block Test (BBT) the patient will be instructed to move as many blocks as possible from one side of the box to the other in 60 seconds, placing only one block at a time. The score obtained is equal to the number of blocks transported in one partition in one minute. It is assessed that the more blocks transported within the established time, the better the manual dexterity of the patient.
Upper limb function and participation - Jebsen Manual Function Test (JTT) | The tests will be applied at pre (baseline), through study completion, an average of 1 month.
  Jebsen Manual Function Test (JTT) will require to the participant to perform six tasks: turning cards and small common objects, simulating feeding, stacking chips, moving large light and heavy objects. Each task will be timed, and the participant will have a maximum of 120 seconds to complete each task.
Upper limb function and participation - Fugl-Meyer Assessment Scale | The tests will be applied at pre (baseline), through study completion, an average of 1 month.
  Fugl-Meyer Assessment Scale will be used to measure range of motion, coordination, reflex activity, tactile sensitivity, and proprioception of the shoulder, elbow, wrist, and hand regions. The scale can be divided into two domains: motor (66 points) and sensory (12). The scoring can be from zero to three points, where: absent function is 0, 1 (one) is partial function, and 2 (two) is normal function. The minimally clinically important difference of this scale is 10% of the gross value, which is 6.6 points in the motor domain and 1.2 points in the sensory domain. Only scores for the affected limb will be considered.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Tecnológica Federal do Paraná, Curitiba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No
Ethical or Consent Restrictions: Participants may not have given explicit consent for their data to be shared beyond the original study.
  Legal or Institutional Policies: Data sharing may be restricted by Brazillian laws.

REFERENCES:
- [Background] Liu M, Xu L, Li H, Chen S, Chen B. Morphological and Functional Changes of the Tibialis Anterior Muscle After Combined Mirror Visual Feedback and Electromyographic Biofeedback in Poststroke Patients: A Randomized Trial. Am J Phys Med Rehabil. 2021 Aug 1;100(8):766-773. doi: 10.1097/PHM.0000000000001628. PMID 33105154
- [Background] Nordio S, Arcara G, Berta G, Dellai A, Brisotto C, Koch I, Cazzador D, Aspidistria M, Ventura L, Turolla A, D'Imperio D, Battel I. Biofeedback as an Adjunctive Treatment for Post-stroke Dysphagia: A Pilot-Randomized Controlled Trial. Dysphagia. 2022 Oct;37(5):1207-1216. doi: 10.1007/s00455-021-10385-2. Epub 2021 Nov 12. PMID 34767083
- [Background] Hou M, Zhao Y, Zhao L, Yuan X, Liu Z, Li H. Efficacy of game training combined with surface electromyography biofeedback on post-stroke dysphagia. Geriatr Nurs. 2024 Jan-Feb;55:255-262. doi: 10.1016/j.gerinurse.2023.11.019. Epub 2023 Dec 12. PMID 38091711
- [Background] Winstein CJ, Stein J, Arena R, Bates B, Cherney LR, Cramer SC, Deruyter F, Eng JJ, Fisher B, Harvey RL, Lang CE, MacKay-Lyons M, Ottenbacher KJ, Pugh S, Reeves MJ, Richards LG, Stiers W, Zorowitz RD; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Quality of Care and Outcomes Research. Guidelines for Adult Stroke Rehabilitation and Recovery: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2016 Jun;47(6):e98-e169. doi: 10.1161/STR.0000000000000098. Epub 2016 May 4. PMID 27145936
- [Background] Feng S, Tang M, Huang G, Wang J, He S, Liu D, Gu L. EMG biofeedback combined with rehabilitation training may be the best physical therapy for improving upper limb motor function and relieving pain in patients with the post-stroke shoulder-hand syndrome: A Bayesian network meta-analysis. Front Neurol. 2023 Jan 10;13:1056156. doi: 10.3389/fneur.2022.1056156. eCollection 2022. PMID 36703623
- [Background] Woodford H, Price C. EMG biofeedback for the recovery of motor function after stroke. Cochrane Database Syst Rev. 2007 Apr 18;2007(2):CD004585. doi: 10.1002/14651858.CD004585.pub2. PMID 17443550
- [Background] Elshafey MA, Abd-Elaziem A, Gouda RE. Functional stretching exercise submitted for spastic diplegic children: a randomized control study. Rehabil Res Pract. 2014;2014:814279. doi: 10.1155/2014/814279. Epub 2014 Jul 20. PMID 25143834
- [Background] Koh SH, Park HH. Neurogenesis in Stroke Recovery. Transl Stroke Res. 2017 Feb;8(1):3-13. doi: 10.1007/s12975-016-0460-z. Epub 2016 Mar 18. PMID 26987852